CLINICAL TRIAL: NCT04956224
Title: A Phase III, Open Label, Multicenter, Single Arm Study to Assess the Safety, Tolerability and Immunogenicity of VLA2001 in Volunteers Aged ≥ 56 Years.
Brief Title: Safety and Immunogenicity of VLA2001 Adults Aged ≥56 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VLA2001-304
Record Dates: First submitted 2021-06-21; First posted 2021-07-09 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: SARS-CoV-2 Virus Infection
Keywords: VLA2001; SARS-CoV-2 Virus Infection; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — VLA2001 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VLA2001 (Experimental)
  Interventions: Biological: VLA2001

INTERVENTIONS:
Biological: VLA2001 — whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG) 1018 in combination with aluminium hydroxide (Wuhan strain)
  2 vaccinations 28 days apart
  Booster Vaccination on Visit B1

SUMMARY:
This is a A Phase III, Open label, Multicenter, Single Arm Study to assess the Safety, Tolerability and Immunogenicity of VLA2001 in volunteers aged ≥ 56 years. Approximately 300 participants are enrolled in a non-randomized manner.

DETAILED DESCRIPTION:
This Phase 3 study is designed as a Multicentre, Open Label, Single Arm Study to assess the Safety, Tolerability and Immunogenicity of VLA2001.

Participants aged 56 years or older and who are either generally healthy or are with a stable medical condition are enrolled.

Approximately 300 participants will be enrolled in a non-randomized manner to receive VLA2001 at the recommended dose level, 28 days apart on Days 1 and 29.

Immunogenicity and safety will be assessed up to month 12 after the first vaccination.

All participants, except those who already received a licensed COVID-19 vaccine outside of the study, will be offered a booster dose with VLA2001. All eligible and willing participants will receive a booster vaccination with VLA2001 and will have a follow-up visit 14 days after the booster dose. The participants will have 1 more follow-up visit 6 months after the booster vaccination which replaces Day 365 for those participants who received a booster dose.

This study will support the VLA2001 safety and immunogenicity database for vaccines aged ≥56 years.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must have read, understood, and signed the informed consent form (ICF).
2. Participants of either gender aged 56 years or older at screening.
3. Medically stable such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain on study through the end of protocol-specified follow-up.
4. Participant has a Body Mass Index (BMI) of 18.0-35.0 kg/m2, inclusive, at screening (Visit 0).
5. Must be able to attend all visits of the study and comply with all study procedures, including daily completion of the e-diary for 7 days following each vaccination.
6. Women of childbearing potential (WOCBP), who are sexually active with a man, must be able and willing to use at least 1 highly effective method of contraception (i.e. implant contraceptive, intra-uterine device (IUD) containing either copper or levonorgestrel, male sterilization [vasectomy], female sterilization, injectable contraceptive, oral contraceptive pill, vaginal contraceptive ring, barrier type of birth control measure) from study start until a minimum of 3 months after the last dose of study vaccine (i.e. 3 months after second dose or 3 months after booster dose).
7. WOCBPs must have a negative pregnancy test prior to each vaccination.

Exclusion Criteria:

1. Participant is pregnant or planning to become pregnant within 3 months after last study vaccine administration.
2. History of allergy to any component of the vaccine.
3. History of laboratory-confirmed SARS-CoV infection
4. Participant had close contact to persons with confirmed SARS-CoV-2 infection within 30 days prior to screening.
5. Participant has participated in a clinical study involving an investigational SARS-CoV-2 vaccine or has received or plans to receive a licensed SARS-CoV-2 vaccine during the duration of the study.
6. Significant infection (e.g. positive SARS-CoV-2 RT-PCR) or other acute illness, including fever > 100 °F (> 37.8 °C) 48 hours before vaccination.
7. Participant has a known or suspected defect of the immune system, such as participants with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to the expected day of randomization.
8. Participant has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the participant may be enrolled.
9. History of drug dependency or current use of drug of abuse or alcohol abuse at screening.
10. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to the expected day of first vaccination or the booster administration.
11. History of clinically significant bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
12. Severe and uncontrolled ongoing autoimmune or inflammatory disease, history of Guillain-Barre syndrome or any other demyelinating condition.
13. Any other significant disease, disorder or finding which in the opinion of the investigator may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study.

    Prior/concomitant therapy:
14. Receipt of immunoglobulin or another blood product within the 3 months before expected day of first vaccination or the booster administration in this study or those who expect to receive immunoglobulin or another blood product during this study.
15. Receipt of medications and or vaccinations intended to prevent COVID-19.
16. Receipt of any vaccine (licensed or investigational), other than licensed influenza vaccine or for medical emergencies such as tetanus or rabies exporsure, within 28 days prior to the expected day of randomization.

    Others:
17. Any member of the study team or sponsor.
18. An immediate family member or household member of the study's personnel.

Booster Vaccination in participants 56 years and older:

In addition to the above described eligibility criteria, the following criteria must be met:

1. Participant has not received a licensed COVID-19 vaccine during his/her participation in the study.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of any Adverse Events (AE) up to Day 43 post-vaccination | Day 43
Immune response as determined by the geometric mean titer (GMT) of SARS-CoV-2-specific neutralizing antibodies | Day 43
Immune response as determined by the seroconversion rate (SCR) of SARS-CoV-2-specific neutralizing antibodies | Day 43

SECONDARY OUTCOMES:
Frequency and severity of solicited injection site and systemic reactions after each vaccination | within 7 days
Frequency and severity of any unsolicited Adverse Event (AE) | until Day 43
Frequency and severity of any unsolicited vaccine-related Adverse Event (AE) | until Day 43
Frequency and severity of any Serious Adverse Event (SAE) | until Day 365
Frequency and severity of any Adverse Event of Special Interest (AESI) | until Day 365
Proportion of participants with Seroconversion after receipt of 2 doses of study vaccination in terms of SARS-CoV-2-specific neutralizing antibodies | on Day 29, Day 57, Day 71 and Day 208
Immune response as determined by the Geometric Mean Titer (GMT) of SARS-CoV-2-specific neutralizing antibodies | on Day 29, Day 57, Day 71 and Day 208
Proportion of participants with Seroconversion after receipt of 2 doses of study vaccination in terms of S-protein binding IgG levels | on Day 29, Day 57, Day 71 and Day 208
Immune response as determined by the Geometric Mean Titer (GMT) of IgG antibodies to SARS-CoV-2 S-protein | on Day 29, Day 57, Day 71 and Day 208
Geometric Mean Fold Increase (GMFI) of neutralizing antibody (for binding and neutralizing antibodies) | on Day 29, Day 43, Day 57, Day 71 and Day 208
Assessment of T-cell responses from Peripheral Blood Mononuclear Cell (PBMCs) in a subset of participants after in vitro stimulation with SARS-CoV-2 antigens using e.g. ELISpot or intracellular cytokine staining. | on Day 1, Day 43, Day 208, Day 365
Frequency and severity of solicited injection site and systemic reactions | within 7 days after booster vaccination
Frequency and severity of any unsolicited AE (Adverse Event) | up to 6 months after booster vaccination
Frequency and severity of any vaccine-related unsolicited AE (Adverse Event) | up to 6 months after booster vaccination
Frequency and severity of any SAE (Serious Adverse Event) | up to 6 months after booster vaccination
Frequency and severity of any AESI (Adverse Event of Special Interest) | up to 6 months after booster vaccination
Geometric mean fold rise (GMFR) with regards to SARS-CoV-2-specific neutralizing antibodies | from day of booster vaccination up to 14 days after
Geometric Mean Titer (GMT) of SARS-CoV-2 specific neutralizing antibodies including formal non-inferiority testing on the GMT ratio for the booster subgroup who had received 2 doses of VLA2001 for primary immunization | on Day 43 and 14 days after booster vaccination
Proportion of participants with 4-fold increase with regards to SARS-CoV-2-specific neutralizing antibodies | from day of booster vaccination up to 14 days after
Geometric mean fold rise (GMFR) with regards to S-protein binding antibodies | from day of booster vaccination up to 14 days after
Proportion of participants with 4-fold increase with regards to S-protein binding antibodies | from day of booster vaccination up to 14 days after
Geometric Mean Titer (GMT) measured as IgG antibodies against SARS-CoV-2 as determined by ELISA | from day of booster vaccination up to 6 months after
Assessment of T-cell responses from Peripheral Blood Mononuclear Cell (PBMCs) in participants after in vitro stimulation with SARS-CoV-2 antigens using ELISpot | from day of booster vaccination up to 6 months after

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Deveopment, Study Chair — Valneva Austria GmbH
Locations (8):
- New Zealand (8):
  - Southern Clinical Trials Waitemata, Auckland, Birkenhead
  - Lakeland Clinical Trials Waikato, Hamilton, Nawton
  - Southern Clinical Trials Totara, Auckland, New Lynn
  - Lakeland Clinical Trials Culloden, Papamoa, Papamoa Beach
  - Southern Clinical Trials Remuera, Auckland, Remuera
  - Southern Clinical Trials Tasman, Nelson, Stoke
  - Southern Clinical Trials Christchurch, Christchurch
  - Lakeland Clinical Trials Rotorua, Rotorua

IPD SHARING:
Plan to Share IPD: No